CLINICAL TRIAL: NCT01308671
Title: Influence of Varenicline on the Antiplatelet Action of Clopidogrel : the Randomized, Open-label VACL (Varenicline Clopidogrel) Study
Brief Title: Influence of Varenicline on the Antiplatelet Action of Clopidogrel
Acronym: VACL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: General Hospital of Chinese Armed Police Forces (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCTC-001-WS704502
Record Dates: First submitted 2011-01-28; First posted 2011-03-04 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-04

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; varenicline; clopidogrel
MeSH Terms: conditions — Coronary Artery Disease | interventions — Varenicline; Counseling; Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- varenicline (Active Comparator): On 3 day after received clopidogrel 75mg/day, Varenicline group will be administered with varenicline 0.5mg Qd,after 3 days, 0.5mg Bid,after 7days,1mg Bid .And received counseling and psychosocial support.
  Interventions: Drug: Varenicline; Behavioral: Counseling and psychosocial support
- Blank (Other): Blank group will be only administered with Counseling and psychosocial support,beside antiplatelet etc.conventional therapy for 14 days.
  Interventions: Behavioral: Counseling and psychosocial support

INTERVENTIONS:
Drug: Varenicline — Varenicline will be administrated 0.5 mg Qd for 3 days,0.5 mg Bid for 4 days, and then 1 mg Bid for 14 days
  Other Names: Champix
  Arms: varenicline
Behavioral: Counseling and psychosocial support — Blank group will receive the same counseling and psychosocial support as varenicline group
  Other Names: nonpharmacologic therapy

SUMMARY:
The purpose of this study is to investigate the effects of steady-state varenicline on the antiplatelet action of clopidogrel in patients with coronary artery disease.

DETAILED DESCRIPTION:
Smoking is a major risk factor for cardiovascular disease (CVD). Compared with nonsmokers, smokers are approximately twice as likely to develop CVD, and three times more likely to die from it. This increased risk is due to the deleterious effects of smoking on endothelial function and blood coagulation, and the development of coronary atherosclerotic plaques. A research showed that continued smoking after successful percutaneous coronary intervention(PCI) is associated with an increased risk of restenosis. However, smoking cessation can make a 36% reduction in crude relative risk (RR) of mortality for patients with CVD. Hence current management guidelines now advocate smoking cessation, in addition to controlling hypertension and dyslipidemia, as part of an overall cardiovascular risk reduction strategy. Varenicline is a novel selective nicotinic acetylcholine receptor partial agonist that has been approved in over 70 countries worldwide as an aid to smoking cessation. Clopidogrel is widely used by patients with coronary artery disease undergoing PCI. The relationship between smoking and cardiovascular disease increases the prospect of patients receiving smoking cessation therapy and Clopidogrel concomitantly in clinical practice. Plasma protein binding of Varenicline is low(≤20%) and independent of age or renal function. The major route of clearance for varenicline is renal excretion. Clopidogrel, a prodrug, is metabolized by 2 consecutive cytochrome P450-dependent steps to its active metabolite, which binds irreversibly to the platelet P2Y12 receptor. The likelihood of a clinically relevant drug-drug interaction between varenicline and Clopidogrel was considered to be low; nevertheless, the possibility of an interaction between these 2 drugs is lack of clinical evidences. Hence, our hypothesis is that varenicline may have no influence on the antiplatelet action of clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

* patients with coronary artery disease(CAD) undergoing PCI in hospital
* smoke 10 or more cigarettes per day
* fewer than 3 months of smoking abstinence in the past year
* motivation to stop smoking

Exclusion Criteria:

* history of previous treatment with clopidogrel or varenicline
* thrombocytopenia(<150,000 platelets/ml)
* bleeding disorder
* liver disease
* gastrointestinal ulcer
* pregnancy
* cancer
* clinically significant allergic reactions
* mental disorders
* drug or alcohol abuse

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2010-10; Primary Completion 2015-12 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
The platelet reactivity index (PRI) values in the two groups | 14 days
  To compare PRI values at the 14-day-treatment period between the 2 groups.

SECONDARY OUTCOMES:
Platelet aggregometry values in the two groups | 7days,14 days
  To compare platelet aggregometry values at the 7-day,14-day-treatment period between the 2 groups.
Urea nitrogen （BUN） and creatinine（Cr）values in the two groups | 7days, 14 days
  To compare BUN and Cr values at the 7-day,14-day-treatment period between the 2 groups.
Number of patients with adverse events and serious adverse events as a measure of safety in the two groups | 7 days,14 days
  To compare the number of patients with adverse events and serious adverse events at the 7-day,14-day-treatment period between the 2 groups

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liang Liu, Doctor, Principal Investigator — Department of Cardiology of General Hospital of Chinese People's Armed Police Forces
Locations (1):
- General Hospital of Chinese People's Armed Police Forces, Beijing, China

REFERENCES:
- [Result] Puranik R, Celermajer DS. Smoking and endothelial function. Prog Cardiovasc Dis. 2003 May-Jun;45(6):443-58. doi: 10.1053/pcad.2003.YPCAD13. PMID 12800127
- [Result] Sojka JE, Weiss JS, Samuels ML, You GM. Effect of the somatostatin analogue octreotide on gastric fluid pH in ponies. Am J Vet Res. 1992 Oct;53(10):1818-21. PMID 1456527
- [Result] McGill HC Jr, McMahan CA, Malcom GT, Oalmann MC, Strong JP. Effects of serum lipoproteins and smoking on atherosclerosis in young men and women. The PDAY Research Group. Pathobiological Determinants of Atherosclerosis in Youth. Arterioscler Thromb Vasc Biol. 1997 Jan;17(1):95-106. doi: 10.1161/01.atv.17.1.95. PMID 9012643
- [Result] Galan KM, Deligonul U, Kern MJ, Chaitman BR, Vandormael MG. Increased frequency of restenosis in patients continuing to smoke cigarettes after percutaneous transluminal coronary angioplasty. Am J Cardiol. 1988 Feb 1;61(4):260-3. doi: 10.1016/0002-9149(88)90927-7. PMID 2963518
- [Result] Critchley JA, Capewell S. Mortality risk reduction associated with smoking cessation in patients with coronary heart disease: a systematic review. JAMA. 2003 Jul 2;290(1):86-97. doi: 10.1001/jama.290.1.86. PMID 12837716
- [Result] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; National Heart, Lung, and Blood Institute Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure; National High Blood Pressure Education Program Coordinating Committee. The Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure: the JNC 7 report. JAMA. 2003 May 21;289(19):2560-72. doi: 10.1001/jama.289.19.2560. Epub 2003 May 14. PMID 12748199
- [Result] Obach RS, Reed-Hagen AE, Krueger SS, Obach BJ, O'Connell TN, Zandi KS, Miller S, Coe JW. Metabolism and disposition of varenicline, a selective alpha4beta2 acetylcholine receptor partial agonist, in vivo and in vitro. Drug Metab Dispos. 2006 Jan;34(1):121-30. doi: 10.1124/dmd.105.006767. Epub 2005 Oct 12. PMID 16221753
- [Result] Burstein AH, Clark DJ, O'Gorman M, Willavize SA, Brayman TG, Grover GS, Walsky RL, Obach RS, Faessel HM. Lack of pharmacokinetic and pharmacodynamic interactions between a smoking cessation therapy, varenicline, and warfarin: an in vivo and in vitro study. J Clin Pharmacol. 2007 Nov;47(11):1421-9. doi: 10.1177/0091270007307574. PMID 17962429
- [Result] Bliden KP, Dichiara J, Lawal L, Singla A, Antonino MJ, Baker BA, Bailey WL, Tantry US, Gurbel PA. The association of cigarette smoking with enhanced platelet inhibition by clopidogrel. J Am Coll Cardiol. 2008 Aug 12;52(7):531-3. doi: 10.1016/j.jacc.2008.04.045. PMID 18687246
- [Result] Schwarz UR, Geiger J, Walter U, Eigenthaler M. Flow cytometry analysis of intracellular VASP phosphorylation for the assessment of activating and inhibitory signal transduction pathways in human platelets--definition and detection of ticlopidine/clopidogrel effects. Thromb Haemost. 1999 Sep;82(3):1145-52. PMID 10494779
- [Result] Aleil B, Ravanat C, Cazenave JP, Rochoux G, Heitz A, Gachet C. Flow cytometric analysis of intraplatelet VASP phosphorylation for the detection of clopidogrel resistance in patients with ischemic cardiovascular diseases. J Thromb Haemost. 2005 Jan;3(1):85-92. doi: 10.1111/j.1538-7836.2004.01063.x. PMID 15634270